CLINICAL TRIAL: NCT01624675
Title: A Double-blind, Placebo-controlled Study, Followed by an Open-label Extension Study Evaluating the Efficacy and Safety of Risperidone (R064766) in Children and Adolescents With Irritability Associated With Autistic Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Risperidone (R064766) in Children and Adolescents With Irritability Associated With Autistic Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100877; RIS-AUT-JPN-01 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Autistic Disorder in Children and Adolescents
Keywords: Autistic disorder in children and adolescents; Risperidone (R064766); Children; Adolescents; Irritability; Autistic disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Risperidone (Experimental): Subjects weighing less than 20 kilogram (kg) received risperidone 0.25 milligram per day (mg/day) up to Day 4. On Day 4, dose was titrated in increments of 0.25 mg/day (up to a daily dose of 1.0 mg) at the regular study visit thereafter till Week 8. Subjects weighing greater than or equal to (>=) 20 kg received risperidone 0.5 mg/day up to Day 4. On Day 4, dose was titrated in increments of 0.5 mg per day (up to a daily dose of 2.5 mg) at the regular visit thereafter till Week 8. The maximum daily dose for subjects weighing >= 45 kg was 3.0 mg. For subjects weighing >=45 kg, the maximum daily dose was 3.0 mg.
  Interventions: Drug: Risperidone
- Placebo (Placebo Comparator): Subjects will receive placebo matching with risperidone orally up to 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — Subjects weighing less than 20 kilogram (kg) received risperidone 0.25 milligram per day (mg/day) up to Day 4. On Day 4, dose was titrated in increments of 0.25 mg/day (up to a daily dose of 1.0 mg) at the regular study visit thereafter till Week 8. Subjects weighing greater than or equal to (>=) 20 kg received risperidone 0.5 mg/day up to Day 4. On Day 4, dose was titrated in increments of 0.5 mg per day (up to a daily dose of 2.5 mg) at the regular visit thereafter till Week 8. The maximum daily dose for subjects weighing >= 45 kg was 3.0 mg. For subjects weighing >=45 kg, the maximum daily dose was 3.0 mg.
  Arms: Risperidone
Drug: Placebo — Subjects will receive placebo matching with risperidone orally up to 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of risperidone compared with placebo in children and adolescents with irritability associated with autistic disorder.

DETAILED DESCRIPTION:
This is a randomized (the drug is assigned by chance), 8-week, double-blind (neither physician nor patient knows the treatment that the patient receives), placebo-controlled (placebo is an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), parallel-group (each group of patients will be treated at the same time), flexible-dose, multicenter study. It will be followed by a 48-week, flexible-dose, open-label (all people know the identity of the intervention) extension, to evaluate the efficacy and safety of risperidone in children and adolescents with a diagnosis of autistic disorder (severe form of pervasive developmental disorder) who have associated irritability. The study consists of up to 2-week screening phase, an 8-week double-blind phase, a 48-week open-label phase, and a 1-week follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic for autistic disorder
* A Clinical Global Impression - Severity (CGI-S) score of =>4 and an Aberrant Behavior Checklist - Japanese Version (ABC-J) Irritability Subscale score of =>18
* Patients with mental age of >18 months as measured by appropriate developmental or mental scales
* Patients who have an appropriate caregiver, eg, parent or study-site personnel, who is able to observe the patient's condition, provide information, and evaluate the patient's response appropriately

Exclusion Criteria:

* Patients with previous or current psychotic disorder (eg, schizophrenia, bipolar disorder, or other psychiatric disorders) or with pervasive developmental disorder not otherwise specified, Asperger's disorder, Rett's disorder, pediatric destructive behavior disorder, or substance dependence
* Patients with a clinically significant endocrine, metabolic, cardiac, hepatic, renal, or pulmonary disorder, or hypertension
* Weight of <15 kg at the time of screening and baseline
* Patients with QTc>450 msec in the standard 12-lead electrocardiogram (ECG) at the time of screening
* Patients with known hypersensitivity to risperidone or paliperidone

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2012-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The change from baseline in the Aberrant Behavior Checklist-Japanese Version (ABC-J) Irritability Subscale scores | Baseline, Week 8
  The ABC-J Irritability subscale consists of 15 items. Each item scores range from 0 to 3: 0 = No problem, 1 = Mild aberrant behavior, 2 = Moderate aberrant behavior, and 3 = Severe aberrant behavior. Higher scores represent worse condition.

SECONDARY OUTCOMES:
The changes from baseline in the subscale scores of Aberrant Behavior Checklist-Japanese Version (ABC-J) at each evaluation of the double-blind phase | Baseline, Week 2, Week 4, Week 6
  The ABC-J consists of 58 items divided into 5 subscales: Irritability, Lethargy and Social withdrawal, Stereotypic behavior, Hyperactivity/Noncompliance, and Inappropriate speech. Each item scores range from 0 to 3: 0 = No problem, 1 = Mild aberrant behavior, 2 = Moderate aberrant behavior, and 3 = Severe aberrant behavior. Higher scores represent worse condition.
The changes from baseline in the subscale scores of Aberrant Behavior Checklist-Japanese Version (ABC-J) at each evaluation of the open-label phase | Baseline, Week 2, Week 4, Week 8, Week 16, Week 24, Week 32, Week 40, Week 48
  The ABC-J consists of 58 items divided into 5 subscales: Irritability, Lethargy and Social withdrawal, Stereotypic behavior, Hyperactivity/Noncompliance, and Inappropriate speech. Each item scores range from 0 to 3: 0 = No problem, 1 = Mild aberrant behavior, 2 = Moderate aberrant behavior, and 3 = Severe aberrant behavior. Higher scores represent worse condition.
The changes from baseline in scores of the Clinical Global Impression - Severity (CGI-S) at each evaluation time point of the double-blind phase | Baseline, Week 1, Week 2, Week 3, Week 4, Week 6, Week 8
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients". Higher scores indicate worsening.
The changes from baseline in scores of the Clinical Global Impression - Severity (CGI-S) at each evaluation time point of the open-label-phase | Baseline, Week 1, Week 2, Week 3, Week 4, Week 8, Week 16, Week 24, Week 32, Week 40, Week 48
  The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a patient. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill patients". Higher scores indicate worsening.
The changes from baseline in scores of the Children's Global Assessment Scale (C-GAS) at each evaluation time point of the double-blind phase and open-label-phase | Baseline, Week 4, Week 8
  The C-GAS rates the patient's general psychological and social functioning on scores ranging from 1 through 100. Lower scores (range 1-10) mean that the patient needs constant supervision; higher scores (range 91-100) mean that the patient has a superior functioning in all areas.
The changes from baseline in scores of the Children's Global Assessment Scale (C-GAS) at each evaluation time point of open-label-phase | Baseline, Week 4, Week 8, Week 16, Week 24, Week 32, Week 40, Week 48
  The C-GAS rates the patient's general psychological and social functioning on scores ranging from 1 through 100. Lower scores (range 1-10) mean that the patient needs constant supervision; higher scores (range 91-100) mean that the patient has a superior functioning in all areas.
The Clinical Global Impression-Change (CGI-C) at each evaluation time point of the double-blind phase | Week 1, Week 2, Week 3, Week 4, Week 6, Week 8
  The CGI-C assesses the patient's condition on the basis of the rater's impression, on a 7-point scale ranging from 1 (Very much improved) to 7 (Very much worse).
The Clinical Global Impression-Change (CGI-C) at each evaluation time point of the open label-phase | Week 1, Week 2, Week 3, Week 4, Week 8, Week 16, Week 24, Week 32, Week 40, Week 48
  The CGI-C assesses the patient's condition on the basis of the rater's impression, on a 7-point scale ranging from 1 (Very much improved) to 7 (Very much worse).
The Parent Satisfaction Questionnaire (PSQ) at each evaluation time point of the double-blind phase | Week 1, Week 2, Week 3, Week 4, Week 6, Week 8
  The PSQ evaluates the caregiver's satisfaction with the study drug.
The Parent Satisfaction Questionnaire (PSQ) at each evaluation time point of the open label-phase | Week 1, Week 2, Week 3, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Week 28, Week 32, Week 36, Week 40, Week 44, Week 48
  The PSQ evaluates the caregiver's satisfaction with the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (17):
- Japan (17):
  - Fuchū
  - Fukui
  - Hirakata
  - Ichikawa
  - Kanzaki
  - Kobe
  - Kodaira
  - Kurashiki
  - Neyagawa
  - Okayama
  - Sakai
  - Shimotsuke
  - Tokyo
  - Toyama
  - Tsu
  - Tsuyama
  - Yokohama

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- See also: A Double-blind, Placebo-controlled Study, Followed by an Open-label Extension Study Evaluating the Efficacy and Safety of Risperidone (R064766) in Children and Adolescents with Irritability Associated with Autistic Disorder — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=3545&filename=CR100877_CSR.pdf